CLINICAL TRIAL: NCT03115788
Title: The Effect of Pain on Short Term Cognitive Performance Using a Computer Assisted/Ipad Game Interface
Brief Title: Pain Effect on Attention Using an Ipad Game App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00037185
Record Dates: First submitted 2017-01-23; First posted 2017-04-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Function
Keywords: Thermal; ipad; game

STUDY DESIGN:
Intervention Model Description: 2 groups; control and treated
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention Game play (Active Comparator): The person will be instructed how to hold the iPad and how to play the game.
  Interventions: Other: iPad
- Thermal pain and ipad performance (Experimental): Interventions: Cold induced pain and heat induced pain. The whole group gets thermal heat (n=40) and half (n=20) get cold water foot immersion and half (n=20) get body temperature foot emersion. The person will be instructed how to hold the iPad and how to play the game. The person will then be allowed to play the game until the number of trials is completed or until the person no longer wishes to play.
  Interventions: Other: Heat induced pain; Other: Cold Induced Pain; Other: iPad

INTERVENTIONS:
Other: Heat induced pain — For the heat induced thermal pain, the research nurse will train the subject to estimate pain quantitatively using a 2 cm 2 Peltier controlled thermode (TSA®) applied to the skin of the arm. Typically, the subject is exposed to temperatures between 41° and 49° C using a random staircase method. After the volunteer learns to qualitatively estimate the thermal pain, pain will be established by heating the the leg with a 4 cm2 Peltier controlled thermode (TSA®) for 90 seconds with the probe clamped at a thermal intensity of 47°C.
  Arms: Thermal pain and ipad performance
Other: Cold Induced Pain — Cold pain will be induced by placing a foot in a container of circulating water maintained at 10°C for 90 seconds (n=20). Half (n=20) of the subjects will have the foot placed in body temperature water of 38°C.
  Arms: Thermal pain and ipad performance
Other: iPad

SUMMARY:
Cognitive performance will be studied over time using an iPad game interface called the nine choice human game (5CH) in normal volunteer subjects before during and after experimentally induced thermal (cold or warm) pain or control (no intervention).

DETAILED DESCRIPTION:
Purpose: to assess the effects of pain on performance in a computer game interface of attention and memory and reliability of the repeated testing.

Rationale: The perioperative period may alter the ability to play an iPad game through changes in attention or memory as result of surgery, anesthesia, pain or medications. This study will describe and quantify and isolate any short term reduction in ability to focus and pay attention to the presence of thermal (cold or warm) pain.

Objectives: Determine if cognitive function is altered from thermal pain (cold or warm) using simple computer/ipad games of attentional performance and cognitive function.

Design and Outcomes: In group 1: no interventions will be used and the subjects will play the ipad game at baseline, 5 minutes later and 10 minutes later. In group 2: The subjects will play the ipad game, then 5 minutes later a thermal probe at 47 degrees C for 90 seconds on the arm or leg will be used while the game is being played. Following 10 minutes of recovery, the subject will play the game again, 5 minutes later the subject will have the foot placed in 10 degree water bath or body temperature water bath while the game is played, and the game will be played 10 minutes later after the foot is warm and dry. Visual analog scale (VAS) pain score from 0-10 will be used to assess discomfort. The subject will be able to stop the game or withdraw at any point. The primary outcome measures will be median cue duration (MCD) in the 9CH game. Secondary outcome measures will be number of correct, incorrect, omissions, time to finish trials, and time to quit for the 9CH. A total of 60 subjects will be studied, 20 subject warm probe/cold water, 20 subjects warm probe/body temperature water, and 20 normal subjects with no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-pregnant female volunteers between the ages of 18-55.

Exclusion Criteria:

* Any reported learning disabilities, psychomotor impairment including diagnosis of ADD/ADHD, seizures, debilitating neurologic disorders (muscular dystrophy, multiple sclerosis, etc.), genetic diseases, heart disease, stroke, or memory deficits; anything that would impair the ability to hold the iPAD and perform the computer gaming tasks (i.e. blindness, color blindness, upper extremity dysfunction or pain). Also any history of cold induced impaired circulation, cold agglutinins or Raynaud's or insensitivity to cold.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Median cue duration | 2 minutes
  ipad game performance

SECONDARY OUTCOMES:
number correct | 2 minutes
  ipad game performance
Premature discontinuation of game | 2 minutes
  ipad game performance
Number of omitted responses | 2 minutes
  ipad game performance

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Ririe, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03115788/ICF_000.pdf